CLINICAL TRIAL: NCT05841290
Title: The Incidence of Postoperative Pain After Using Different Types of Sealers (A Randomized Clinical Trial)
Brief Title: The Incidence of Postoperative Pain After Using Different Types of Sealers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Kareem darwish, Teaching Assistant, Endodontics department , Faculty of dentistry brititsh university in egypt, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-017
Record Dates: First submitted 2022-12-16; First posted 2023-05-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain; Root Canal Sealers; Sillicon Based Sealers; Resin Based Sealers
MeSH Terms: conditions — Pain, Postoperative | interventions — Therapeutic Irrigation; epoxy resin-based root canal sealer; Dental Occlusion; Pain Measurement

STUDY DESIGN:
Intervention Model Description: Root Canal Treatment (RCT) with 2 parallel groups, two arms, superiority trial with 1:1 allocation ratio
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (1) Resin Based Sealer intervention (Experimental): evaluate the incidence and intensity of post-operative pain after obturation using resin based sealers.
  Interventions: Procedure: Primary local anesthesia; Procedure: Supplemental local anesthesia; Procedure: Removal Of Caries and Access Cavity; Procedure: Rubber dam isolation of tooth; Procedure: Bleeding control; Procedure: Canal negotiation; Procedure: Coronal flaring; Procedure: Working Length Determination (W.L); Procedure: Glide path; Procedure: Irrigation; Procedure: Cleaning and shaping using rotary system; Procedure: Second w.l determination; Procedure: Apical gauging; Procedure: Activation of the irrigant; Procedure: Master cone check; Drug: application of resin based sealer inside the canal in the resin based sealer group; Diagnostic Test: application of the sillicon based sealer inside the canal in the sillicon based group; Procedure: Obturation; Diagnostic Test: Visual Analogue Scale (VAS)
- Group (2) Silicone Based Sealer intervention (Experimental): evaluate the incidence and intensity of post-operative pain after obturation using sillicon based sealers.
  Interventions: Procedure: Primary local anesthesia; Procedure: Supplemental local anesthesia; Procedure: Removal Of Caries and Access Cavity; Procedure: Rubber dam isolation of tooth; Procedure: Bleeding control; Procedure: Canal negotiation; Procedure: Coronal flaring; Procedure: Working Length Determination (W.L); Procedure: Glide path; Procedure: Irrigation; Procedure: Cleaning and shaping using rotary system; Procedure: Second w.l determination; Procedure: Apical gauging; Procedure: Activation of the irrigant; Procedure: Master cone check; Drug: application of resin based sealer inside the canal in the resin based sealer group; Diagnostic Test: application of the sillicon based sealer inside the canal in the sillicon based group; Procedure: Obturation; Diagnostic Test: Visual Analogue Scale (VAS)

INTERVENTIONS:
Procedure: Primary local anesthesia — Tooth will be anaesthetized using Local anesthesia containing Articaine with epinephrine 1:100,000.
Procedure: Supplemental local anesthesia — if needed
  Other Names: intraligamentary injection / Intrapulpal Anesthesia
Procedure: Removal Of Caries and Access Cavity — • Access cavity will be performed using a carbide round steel bur and tapered diamond stone until complete deroofing.
Procedure: Rubber dam isolation of tooth — Rubber dam isolation of tooth using certain clamps .
Procedure: Bleeding control — bleeding is controlled by using excavator for the removing the pulp tissue . using a piece of cotton soaked with Sodium hypochlorite. using local anesthesia with vasoconstrictor if needed and if suitable for the patient.
Procedure: Canal negotiation — Coronal patency of the coronal and the Middle part of the canal using file #10 Apical patency of the apical part of the canal using #10
  Other Names: Coronal patency; Apical patency
Procedure: Coronal flaring — Coronal flaring using Orifice opener of a certain Rotary system in and out motion first then brushing motion touching all the canal walls
Procedure: Working Length Determination (W.L) — Working length determination (W.L) using #10 K File , working length is recorded using apex locator and confirmatory radiograph.
Procedure: Glide path — Glide path of the canal Using #10 ,15 ,20 ,25 K files till becoming Super-Loose Inside the Canal at the recorded w.l to create a path for the rotary file .
Procedure: Irrigation — Irrigation using 5.25% sodium hypochlorite introduced using side vented needle
Procedure: Cleaning and shaping using rotary system — Cleaning and shaping using rotary system plus irrigation and apical patency between every rotary file .
Procedure: Second w.l determination — Second w.l determination using electronic apex locator before using final finishing rotary file .
Procedure: Apical gauging — Establish the depth of apical constriction - this is the zero reading on your apex locator. your working length will be 0.5mm - 1mm short of this.
  After cleaning and preparing the canal system to your working length, passively insert 02 taper hand files, starting from #15. If the file goes past the apical constriction (your working length + 0.5-1mm), then choose the next largest file and repeat.
  When a file passively binds short of the apical constriction, that will be the upper limit of the apical constriction diameter. The smaller file before that would be the lower limit.
  Apical gauging helps with:
  Choosing the best master cone that closely matches canal length and taper Achieving true tug back - as opposed to false tug back! Minimising gutta percha extrusions during obturation
Procedure: Activation of the irrigant — Activation of the irrigant using Manual Dynamic Agitation and Ultra x or eddy tips for activation
Procedure: Master cone check — Master cone check Clinically and confirmatory radiograph
Drug: application of resin based sealer inside the canal in the resin based sealer group — application done by inserting inside the canal by spreader or master cone
  Other Names: AH plus
Diagnostic Test: application of the sillicon based sealer inside the canal in the sillicon based group — application done by injection inside the canal
  Other Names: Gutta flow 2
Procedure: Obturation — done by lateral condensation technique
Diagnostic Test: Visual Analogue Scale (VAS) — Pain is evaluated using visual analogue scale (VAS) which is a pain rating scale. Scores are based on measures that are self-reported of symptoms that are recorded through a single handwritten mark placed at one point along the length of a 10-cm line representing a continuum between the two ends of the scale; on the left end of the scale (0 cm) means "no pain" and the on the right end of the scale (10 cm) "worst pain"

SUMMARY:
The aim of this randomized clinical trial is to evaluate and compare the incidence and intensity of post-operative pain after obturation using resin and silicon-based sealers.

DETAILED DESCRIPTION:
The main objectives of root canal therapy are to achieve long-term comfort, function, and aesthetics for the patients and prevention of reinfection of tooth. These objectives are provided through complete cleaning, shaping, and obturation of canals of affected teeth .

Some patients may report moderate-to-severe pain and/or swelling following root canal treatment .

This is detrimental for both patient and dentist and may entail an unscheduled emergency visit by patients to relieve their symptoms.

Postoperative pain is considered a clinical outcome that exhibits the multifactorial nature of patients' responses to variables among treatment procedures such as maintaining the working length to the apical constriction, finishing the endodontic treatment in single visit or multiple visit, instrumentation technique and the type of endodontic sealer used for obturation .

Such pain occurrence is mainly due to mechanical, chemical or microbial injury to the periapical tissues .

Trauma of periapical tissue or bacterial extrusion and root canal sealer specifically, extrusion of root canal sealer can disrupt periodontal tissues and cause inflammatory reactions. The intensity of this reaction depends on the composition of the sealer .

Root canal sealers can play a crucial role in this regard by coming in contact with the periapical tissues through apical foramen and lateral canals causing a localized inflammation with a direct influence on the degree of inflammation based on the composition of the sealer in turn influencing postoperative pain levels .

Silicone is inert and biocompatible and has been widely used in medicine as an implant material Silicone-based root-canal sealers are also available. However, there are no data on the clinical performance of this type of material in endodontic treatment .

ELIGIBILITY:
Inclusion Criteria:

* • Patient's age ranges from 18-50 years old.

  * Patients with teeth diagnosed with symptomatic irreversible pulpitis.
  * Normal periapical condition confirmed by normal periapical radiograph
  * The teeth are restorable
  * Teeth are periodontally free, with no mobility and negative to percussion and palpation test.

Exclusion Criteria:

* • Teeth with immature roots

  * Non restorable teeth
  * Medically compromised patients with systemic complication that would alter the treatment.
  * Necrotic teeth
  * Teeth with apical periodontitis or periapical lesions
  * necrotic Teeth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | after 6 hours of endodontic treatment
  Pain is evaluated using visual analogue scale (VAS) which is a pain rating scale. Scores are based on measures that are self-reported of symptoms that are recorded through a single handwritten mark placed at one point along the length of a 10-cm line representing a continuum between the two ends of the scale; on the left end of the scale (0 cm) means "no pain" and the on the right end of the scale (10 cm) "worst pain" Each Outcome Measure should typically only specify a single time point of assessment
Postoperative pain | after 12 hours of endodontic treatment
  Pain is evaluated using visual analogue scale (VAS) which is a pain rating scale. Scores are based on measures that are self-reported of symptoms that are recorded through a single handwritten mark placed at one point along the length of a 10-cm line representing a continuum between the two ends of the scale; on the left end of the scale (0 cm) means "no pain" and the on the right end of the scale (10 cm) "worst pain"
Postoperative pain | after 24 hours of endodontic treatment
  Pain is evaluated using visual analogue scale (VAS) which is a pain rating scale. Scores are based on measures that are self-reported of symptoms that are recorded through a single handwritten mark placed at one point along the length of a 10-cm line representing a continuum between the two ends of the scale; on the left end of the scale (0 cm) means "no pain" and the on the right end of the scale (10 cm) "worst pain"
Postoperative pain | after 48 hours of endodontic treatment
  Pain is evaluated using visual analogue scale (VAS) which is a pain rating scale. Scores are based on measures that are self-reported of symptoms that are recorded through a single handwritten mark placed at one point along the length of a 10-cm line representing a continuum between the two ends of the scale; on the left end of the scale (0 cm) means "no pain" and the on the right end of the scale (10 cm) "worst pain"
Postoperative pain | after 72 hours of endodontic treatment
  Pain is evaluated using visual analogue scale (VAS) which is a pain rating scale. Scores are based on measures that are self-reported of symptoms that are recorded through a single handwritten mark placed at one point along the length of a 10-cm line representing a continuum between the two ends of the scale; on the left end of the scale (0 cm) means "no pain" and the on the right end of the scale (10 cm) "worst pain"

OTHER OUTCOMES:
sealer extrusion | average 1 week
  The 2 blinded and calibrated examiners will evaluate the immediate periapical radiographs after canal obturation.
  Sealer extrusion will classified to either absent or present.
  If there will be a sealer extrusion in at least 1 root for multirooted teeth, will be regarded as the "presence" of sealer extrusion
  Measured by clinical symptoms and signs ( pain , swelling , parasthesia )
root-filling voids | after obturation is done intra-appointment
  The 2 blinded and calibrated examiners will evaluate the immediate periapical radiographs after canal obturation.
  will classified to either absent or present. If there will be root-filling voids in at least 1 root for multirooted teeth, will be regarded as the "presence" of it
the level of root filling | after obturation is done intra-appointment
  The 2 blinded and calibrated examiners will evaluate the immediate periapical radiographs after canal obturation.
  just discovered it will be corrected

CONTACTS AND LOCATIONS:
Locations (1):
- British University in Egypt, El Shorouk, Cairo Governorate, Egypt

REFERENCES:
- [Background] Torabinejad M, White SN. Endodontic treatment options after unsuccessful initial root canal treatment: Alternatives to single-tooth implants. J Am Dent Assoc. 2016 Mar;147(3):214-20. doi: 10.1016/j.adaj.2015.11.017. Epub 2016 Jan 9. PMID 26778004
- [Background] Javidi M, Zarei M, Ashrafpour E, Gharechahi M, Bagheri H. Post-treatment Flare-up Incidence after Using Nano Zinc Oxide Eugenol Sealer in Mandibular First Molars with Irreversible Pulpitis. J Dent (Shiraz). 2020 Dec;21(4):307-313. doi: 10.30476/DENTJODS.2020.83231.1041. PMID 33344681
- [Background] AlRahabi MK. Predictors, prevention, and management of postoperative pain associated with nonsurgical root canal treatment: A systematic review. J Taibah Univ Med Sci. 2017 May 9;12(5):376-384. doi: 10.1016/j.jtumed.2017.03.004. eCollection 2017 Oct. PMID 31435267
- [Background] Genet JM, Hart AA, Wesselink PR, Thoden van Velzen SK. Preoperative and operative factors associated with pain after the first endodontic visit. Int Endod J. 1987 Mar;20(2):53-64. doi: 10.1111/j.1365-2591.1987.tb00590.x. No abstract available. PMID 3471726
- [Background] Christian Gomes Moura C, Cristina Cunha T, Oliveira Crema V, Dechichi P, Carlos Gabrielli Biffi J. A study on biocompatibility of three endodontic sealers: intensity and duration of tissue irritation. Iran Endod J. 2014 Spring;9(2):137-43. Epub 2014 Mar 8. PMID 24688584
- [Background] Zhang W, Peng B. Tissue reactions after subcutaneous and intraosseous implantation of iRoot SP, MTA and AH Plus. Dent Mater J. 2015;34(6):774-80. doi: 10.4012/dmj.2014-271. PMID 26632225
- [Background] Habal MB. The biologic basis for the clinical application of the silicones. A correlate to their biocompatibility. Arch Surg. 1984 Jul;119(7):843-8. doi: 10.1001/archsurg.1984.01390190081019. PMID 6375634
- [Background] Marcus DA. Interrelationships of neurochemicals, estrogen, and recurring headache. Pain. 1995 Aug;62(2):129-139. doi: 10.1016/0304-3959(95)00052-T. PMID 8545137
- [Background] Dao TT, Knight K, Ton-That V. Modulation of myofascial pain by the reproductive hormones: a preliminary report. J Prosthet Dent. 1998 Jun;79(6):663-70. doi: 10.1016/s0022-3913(98)70073-3. PMID 9627895
- [Background] Walton R, Fouad A. Endodontic interappointment flare-ups: a prospective study of incidence and related factors. J Endod. 1992 Apr;18(4):172-7. doi: 10.1016/S0099-2399(06)81413-5. PMID 1402571
- [Background] Mehrvarzfar P, Shababi B, Sayyad R, Fallahdoost A, Kheradpir K. Effect of supraperiosteal injection of dexamethasone on postoperative pain. Aust Endod J. 2008 Apr;34(1):25-9. doi: 10.1111/j.1747-4477.2007.00076.x. PMID 18352900
- [Background] Ali SG, Mulay S, Palekar A, Sejpal D, Joshi A, Gufran H. Prevalence of and factors affecting post-obturation pain following single visit root canal treatment in Indian population: A prospective, randomized clinical trial. Contemp Clin Dent. 2012 Oct;3(4):459-63. doi: 10.4103/0976-237X.107440. PMID 23633809
- [Background] Watkins CA, Logan HL, Kirchner HL. Anticipated and experienced pain associated with endodontic therapy. J Am Dent Assoc. 2002 Jan;133(1):45-54. doi: 10.14219/jada.archive.2002.0020. PMID 11811742
- [Background] Cleghorn BM, Christie WH, Dong CC. Root and root canal morphology of the human permanent maxillary first molar: a literature review. J Endod. 2006 Sep;32(9):813-21. doi: 10.1016/j.joen.2006.04.014. Epub 2006 Jun 30. PMID 16934622
- [Background] Claffey E, Reader A, Nusstein J, Beck M, Weaver J. Anesthetic efficacy of articaine for inferior alveolar nerve blocks in patients with irreversible pulpitis. J Endod. 2004 Aug;30(8):568-71. doi: 10.1097/01.don.0000125317.21892.8f. PMID 15273637
- [Background] Mikesell P, Nusstein J, Reader A, Beck M, Weaver J. A comparison of articaine and lidocaine for inferior alveolar nerve blocks. J Endod. 2005 Apr;31(4):265-70. doi: 10.1097/01.don.0000140576.36513.cb. PMID 15793381
- [Background] Risso PA, Cunha AJ, Araujo MC, Luiz RR. Postobturation pain and associated factors in adolescent patients undergoing one- and two-visit root canal treatment. J Dent. 2008 Nov;36(11):928-34. doi: 10.1016/j.jdent.2008.07.006. Epub 2008 Sep 3. PMID 18771838
- [Background] Menke ER, Jackson CR, Bagby MD, Tracy TS. The effectiveness of prophylactic etodolac on postendodontic pain. J Endod. 2000 Dec;26(12):712-5. doi: 10.1097/00004770-200012000-00010. PMID 11471639
- [Background] Sathorn C, Parashos P, Messer HH. Effectiveness of single- versus multiple-visit endodontic treatment of teeth with apical periodontitis: a systematic review and meta-analysis. Int Endod J. 2005 Jun;38(6):347-55. doi: 10.1111/j.1365-2591.2005.00955.x. PMID 15910469
- [Background] Spangberg LS. Evidence-based endodontics: the one-visit treatment idea. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Jun;91(6):617-8. doi: 10.1067/moe.2001.116720. No abstract available. PMID 11402269
- [Background] al-Omari MA, Dummer PM. Canal blockage and debris extrusion with eight preparation techniques. J Endod. 1995 Mar;21(3):154-8. doi: 10.1016/s0099-2399(06)80443-7. PMID 7561660
- [Background] Carrotte P. Endodontics: Part 7. Preparing the root canal. Br Dent J. 2004 Nov 27;197(10):603-13. doi: 10.1038/sj.bdj.4811823. PMID 15611742
- [Background] Ng YL, Glennon JP, Setchell DJ, Gulabivala K. Prevalence of and factors affecting post-obturation pain in patients undergoing root canal treatment. Int Endod J. 2004 Jun;37(6):381-91. doi: 10.1111/j.1365-2591.2004.00820.x. PMID 15186245
- [Background] Fonseca B, Coelho MS, Bueno CEDS, Fontana CE, Martin AS, Rocha DGP. Assessment of Extrusion and Postoperative Pain of a Bioceramic and Resin-Based Root Canal Sealer. Eur J Dent. 2019 Jul;13(3):343-348. doi: 10.1055/s-0039-3399457. Epub 2019 Dec 3. PMID 31794999
- [Background] Shim K, Jang YE, Kim Y. Comparison of the Effects of a Bioceramic and Conventional Resin-Based Sealers on Postoperative Pain after Nonsurgical Root Canal Treatment: A Randomized Controlled Clinical Study. Materials (Basel). 2021 May 19;14(10):2661. doi: 10.3390/ma14102661. PMID 34069521
- [Background] Chitra Sachdev Comparative Evaluation of Post-Operative Pain On Unintentional Extruded Three Different Root Canal Sealers Periapically- An Invivo Study. Int J Recent Sci Res. 12(03), pp. 41232-234.
- [Background] Khandelwal A, Jose J, Teja KV, Palanivelu A. Comparative evaluation of postoperative pain and periapical healing after root canal treatment using three different base endodontic sealers - A randomized control clinical trial. J Clin Exp Dent. 2022 Feb 1;14(2):e144-e152. doi: 10.4317/jced.59034. eCollection 2022 Feb. PMID 35173897
- [Background] Alexander I. Electronic medical records for the orthopaedic practice. Clin Orthop Relat Res. 2007 Apr;457:114-9. doi: 10.1097/BLO.0b013e3180342802. PMID 17415063